CLINICAL TRIAL: NCT00785525
Title: Filgrastim-Mobilized Peripheral Blood Stem Cells for Allogeneic Transplantation With Unrelated Donors
Brief Title: Filgrastim-Mobilized Stem Cells for Transplantation Using Unrelated Donors
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PBSC
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy Unrelated Stem Cell Donors
MeSH Terms: interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

INTERVENTIONS:
Drug: Filgrastim — PBSC donors will receive 10 µg/kg of filgrastim subcutaneously each day of a five day mobilization schedule.
  Other Names: Neupogen®, GCSF

SUMMARY:
The purpose of the study is to:

* Establish and evaluate a system for collection of filgrastim-mobilized peripheral blood stem cells from National Marrow Donor Program donors (NMDP) donors
* Assess the safety among NMDP donors of filgrastim administration and PBSC leukapheresis
* Assess the safety and efficacy of filgrastim-mobilized PBSC in unrelated donor hematopoietic stem cell transplant recipients
* Determine the acceptability of stem cell donation by filgrastim stimulated apheresis in normal donors

DETAILED DESCRIPTION:
For many years, allogeneic bone marrow transplantation has been used to successfully treat leukemias, other hematologic conditions and congenital disorders. The first unrelated donor transplants were performed in the late 1970s, but this procedure did not become widely available until the development of several consolidated unrelated donor registries around the world. The National Marrow Donor Program, established in 1987, is the world's largest registry and currently lists more than 7 million donors. Since its beginning, NMDP has facilitated more than 30,000 unrelated transplants.

Although not a licensed indication, considerable experience has been accumulated concerning administration of filgrastim to normal adults. Most of these adults were volunteer research subjects or donors of PBSC for use in related donor transplants. Beginning in February 1997, filgrastim stimulated PBSC have been collected from NMDP donors under protocol. The protocol (locally referred to as G2) began under an NMDP-sponsored Investigational New Drug (IND) application filed with FDA for collecting PBSC for a second donation following an initial donation of bone marrow. In 1999 a second protocol was opened (locally referred to as G1) as requests for PBSC as a primary donation source became more common. In 2005 the two protocols were combined to eliminate redundancy and provide for ease of use.

The protocol establishes and evaluates a system to supply peripheral blood stem cell (PBSC) products for use in unrelated donor hematopoietic stem cell (HSC) transplantation. The protocol describes processes for donor identification, education and evaluation. Procedures for administration and monitoring of the stem cell mobilizing agent filgrastim are included. The protocol also describes procedures for the collection of PBSC products by leukapheresis and includes provisions for long term donor follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. PBSC donors must meet the same criteria as NMDP marrow donors. These criteria are set forth in the Donor Center Manual of Operations.
2. Confirmatory pregnancy test must be performed within 15 days of collection and prior to the start of filgrastim administration; this may require more than one test to be performed.

Exclusion Criteria:

1. Pregnancy or uninterruptible breastfeeding. Pregnancy is an absolute contraindication under this protocol. Women who are breastfeeding must be willing and able to interrupt breastfeeding during the administration of filgrastim and for two days following the final dose.
2. Sensitivity to filgrastim or to E. coli-derived recombinant protein products.
3. History of autoimmune disorders, including rheumatic diseases and thyroid disorders. Exception: As with bone marrow donations, donors with a history of thyroid disease who have undergone successful therapy may be suitable.
4. History of deep vein thrombosis or pulmonary embolism.
5. History of iritis or episcleritis.
6. Thrombocytopenia < 150 x 10^9/L (< 150,000/uL) at baseline evaluation.
7. Current treatment with lithium. Drug interactions between filgrastim and lithium, which may potentiate the release of neutrophils, have not been fully evaluated.
8. Positive Hemoglobin-Solubility (e.g., SickleDex or equivalent) test.
9. Donors receiving experimental therapy or investigational agents.
10. Positive pregnancy test collected/reported prior to start of filgrastim.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60000 (Estimated)
Dates: Start 1997-02 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Establish and evaluate a system for collection of filgrastim-mobilized peripheral blood stem cells from NMDP donors. | Ongoing

SECONDARY OUTCOMES:
Assess the safety among NMDP donors of filgrastim administration and PBSC leukapheresis | Ongoing
Assess the safety and efficacy of filgrastim-mobilized PBSC in unrelated donor hematopoietic stem cell transplant recipients | Ongoing
Determine the acceptability of stem cell donation by filgrastim stimulated apheresis in normal donors | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: John P Miller, MD, PhD, Principal Investigator — National Marrow Donor Program
Locations (4):
- United States (4):
  - Gift of Life Bone Marrow Foundation, Boca Raton, Florida
  - C.W. Bill Young Marrow Donor Center, Rockville, Maryland
  - Be The Match, Minneapolis, Minnesota
  - DKMS Americas, New York, New York

REFERENCES:
- [Derived] Pulsipher MA, Chitphakdithai P, Logan BR, Leitman SF, Anderlini P, Klein JP, Horowitz MM, Miller JP, King RJ, Confer DL. Donor, recipient, and transplant characteristics as risk factors after unrelated donor PBSC transplantation: beneficial effects of higher CD34+ cell dose. Blood. 2009 Sep 24;114(13):2606-16. doi: 10.1182/blood-2009-03-208355. Epub 2009 Jul 16. PMID 19608747
- See also: Donors from this study are drawn from members on the Be The Match Registry who are a possible match for a patient who needs a transplant. If you are interested in becoming a member click on the link and read more about our program. — http://www.marrow.org